CLINICAL TRIAL: NCT04256655
Title: A Phase 1, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of CDX 6114 After Multiple Ascending Oral Dose Administration to Patients With Phenylketonuria (PKU).
Brief Title: Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of CDX 6114 in PKU Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study product composition to move from liquid to solid
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19.05.CLI
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 0.225 g (Experimental): Randomized to treatment with either CDX-6114 0.225g or matching Placebo
  Interventions: Drug: cohort 1 0.225g
- Cohort 2 0.75g (Experimental): Randomized to treatment with either CDX-6114 0.75g or matching Placebo
  Interventions: Drug: Cohort 2 0.75g
- Cohort 3 2.25g (Experimental): Randomized to treatment with either CDX-6114 2.25 g or matching Placebo
  Interventions: Drug: Cohort 3 2.25 g

INTERVENTIONS:
Drug: cohort 1 0.225g — Drug: CDX 6114 CDX-6114 for oral administration is formulated in phosphate buffer, which also includes mannitol and poloxamer.The vehicle solution provided is identical to the CDX-6114 oral solution except for the active drug. Matching Placebo The placebo oral dosing solution will also be supplied as an oral solution and will be made up of the phosphate buffer diluent and the caramel flavoring.
  Other Names: placebo
  Arms: Cohort 1 0.225 g
Drug: Cohort 2 0.75g — Drug: CDX 6114 CDX-6114 for oral administration is formulated in phosphate buffer, which also includes mannitol and poloxamer.The vehicle solution provided is identical to the CDX-6114 oral solution except for the active drug. Matching Placebo The placebo oral dosing solution will also be supplied as an oral solution and will be made up of the phosphate buffer diluent and the caramel flavoring.
  Other Names: placebo
  Arms: Cohort 2 0.75g
Drug: Cohort 3 2.25 g — Drug: CDX 6114 CDX-6114 for oral administration is formulated in phosphate buffer, which also includes mannitol and poloxamer.The vehicle solution provided is identical to the CDX-6114 oral solution except for the active drug. Matching Placebo The placebo oral dosing solution will also be supplied as an oral solution and will be made up of the phosphate buffer diluent and the caramel flavoring.
  Arms: Cohort 3 2.25g

SUMMARY:
The primary objective is of this Phase 1 study is to evaluate the safety and tolerability of daily, multiple, oral doses of CDX-6114 when administered to patients with PKU for 14 days. The aim is to check if administration of daily, multiple, oral doses of CDX-6114 to patients with PKU for 14 days shows a clinically acceptable safety and tolerability profile.

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients between the ages of 18 and 65 years, with a diagnosis of classical PKU
2. Patients with a blood phenylalanine concentration > 600mol/L at screening as an indicator of sub-optimal dietary management
3. Body mass index (BMI) between 18 and 35 kg/m2 at screening.
4. Male patients must agree not to donate sperm starting at screening and continuing throughout the clinical study period up to 90 days after last study drug administration
5. Female patients of childbearing potential and their spouse/partner
6. Female patients of non-childbearing potential:
7. Female patients must agree not to breastfeed. This includes the period starting at screening and continuing throughout the clinical study period up to 90 days after last study drug administration.
8. Female patients must agree not to donate ova. This includes the period starting at screening and continuing throughout the clinical study period up to 90 days after last study drug administration.
9. Patients must be deemed competent to understand the nature of the study and capable of giving written informed consent. Patients must also be willing to attend scheduled study visits in person and to reliably communicate to study personnel on adverse events and concomitant medication use.
10. Patients must agree not to participate in another interventional study while participating in the present clinical study.

Exclusion Criteria

1. Presence or history of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease/condition (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies and childhood asthma).
2. Presence or history of gastrointestinal illness or conditions interfering with normal gastrointestinal anatomy. Examples include gastrointestinal bypass surgery, cholecystectomy, partial or total gastrectomy, gastric band surgery, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or coeliac disease.
3. Active treatment with any platelet aggregation inhibitor and/or active treatment (or within the last 4 weeks) with anticoagulant medication.
4. Presence or history of specific food intolerance. Examples include coeliac disease, severe lactose or dairy food intolerance.
5. Positive result for serum hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (HAV), hepatitis C virus antibodies (HCV), or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of Treatment-Emergent Adverse Events (AEs) will be measured | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat oral administration of CDX-6114 for 14 days assesed by Adverse events monitoring following following repeat-dose, oral administration for 14 days
Change in the serum levels of CDX-6114 will be summarized descriptively over time | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Change in Absolute values and changes from baseline in blood pressure measurements will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by blood pressure monitoring
Change in absolute values and changes from baseline in Respiratory rate measurements will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by respiratory rate monitoring
Change in absolute values and changes from baseline in Heart rate measurements will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Change in absolute values and changes from baseline in body temperature (in Fahrenheit or Celsius) measurements will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by body temperature monitoring
Change in absolute values and changes from baseline in 12 lead Electrocardiogram (ECG) measurements will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by 12 lead ECG including P Wave, QRS Complex, QT Interval
Change in absolute values of Weight measurements will be summarized over time for each treatment using a weighing scale in Kg or pounds over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by weight monitoring
Change in absolute blood composition values from baseline to the last post-dose time-point will be summarized for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by laboratory assessments as Haematology ( routine blood work)
Change in absolute blood composition values from baseline to the last post-dose time-point will be summarized for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by laboratory assessments as Coagulation ( routine blood test)
Change in absolute urine composition values and changes from baseline to the last post-dose time-point will be summarized for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by by routine urinalysis
Any change in the incidence of treatment-Emergent Antibodies will be assesed | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by assessment for development of anti-CDX-6114 antibodies
Change in absolute values of height measurements will be summarized over time for each treatment using length measurement scale in centimeters or inches | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  The safety and tolerability of CDX-6114 following repeat dose oral administration assesed by height examination using Lenght scale

SECONDARY OUTCOMES:
Change in concentration of post parandial plasma level of Phe will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Change in concentration of post parandial plasma level of CA will be summarized over time for each treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Change in the peak Phe concentration in Plasma will be summarized by treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Change in the peak CA concentration in Plasma will be summarized by treatment | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Phe Area under the plasma concentration versus time curve (AUC) , over a 24 hour period, following dosing and the standardized meal | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
CA Area under the plasma concentration versus time curve (AUC) , over a 24 hour period, following dosing and the standardized meal | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Serum concentrations of CDX-6114 over a 24 hour period, following dosing and thestandardized meal | Within 0.25min , 0.5min , 1hours, 2hours, 5hours (immediately prior to starting lunch), 7.5hours, 11.5 hours(immediately prior to starting the evening meal), 14hours and 16 hours after the first dose of study medication on both day 1 and day 14
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points following a repeat dose of CDX-6114 , oral administration for 14 days
Change in attention | The questionnaire will be completed at home by the patient on Day -1 and on Day 13 before each in-house period
  change in attention during the study will be assessed by using the inattention subscale of the Attention-Deficit Hyperactivity Disorder Self-Report Scale (ASRS-v1.1).
Change in mood | The questionnaire will be completed at home by the patient on Day -1 and Day 13 before each in-house period. The POMS-2 questionnaire used is the full-length adult (18+ years) version (POMS 2-A).
  Any change in mood symptoms will be assessed by using the Profile of Mood States 2nd Edition (POMS-2) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Nunes, MD PhD, Study Director — Global Development Lead - GI care